CLINICAL TRIAL: NCT05049798
Title: Assessment of Guselkumab (Tremfya) and IL-17 Inhibitor Therapies in Patients With Psoriatic Arthritis in Routine Clinical Practice; A Prospective, Observational Cohort Study
Brief Title: A Study of Guselkumab and Interleukin-17 (IL-17) Inhibitor Therapies in Participants With Psoriatic Arthritis in Routine Clinical Practice
Acronym: PsABIOnd
Status: Active, not recruiting | Type: Observational
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108938; CNTO1959PSA4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-08-31; First posted 2021-09-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — guselkumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Cohort 1: Guselkumab: Data as available from participant's source medical records will be collected for adult participants with a confirmed diagnosis of Psoriatic Arthritis (PsA) who are starting guselkumab as a first, second, third, or fourth line of PsA biologic therapy either as monotherapy or with other medications per routine clinical practice in main study. Participants who meet the selection criteria for both the main study and substudy, will be consecutively offered to be enrolled into the substudy at the time of enrollment into the main study.
  Interventions: Drug: Guselkumab
- Cohort 2: Interleukin-17 inhibitor (IL-17i): Data as available from participant's source medical records will be collected for adult participants with a confirmed diagnosis of PsA who are starting IL-17i as a first, second, third, or fourth line of PsA biologic therapy either as monotherapy or with other medications per routine clinical practice in main study. Participants who meet the selection criteria for both the main study and substudy, will be consecutively offered to be enrolled into the substudy at the time of enrollment into the main study.
  Interventions: Drug: IL-17i

INTERVENTIONS:
Drug: Guselkumab — Participants will not receive any intervention as a part of this study. Participants who are initiating the treatment with guselkumab, will be observed according to standard clinical practice.
  Other Names: TREMFYA
  Groups: Cohort 1: Guselkumab
Drug: IL-17i — Participants will not receive any intervention as a part of this study. Participants who are initiating the treatment with IL-17i, will be observed according to standard clinical practice.
  Groups: Cohort 2: Interleukin-17 inhibitor (IL-17i)

SUMMARY:
The purpose of this study is to evaluate treatment persistence with guselkumab and interleukin-17 inhibitor (IL-17i) initiated at enrollment into this study (PsABIOnd).

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is a seronegative inflammatory spondylarthritis associated with psoriasis (PsO), which can cause pain and swelling in the joints, sausage-shaped swelling of the fingers and toes (dactylitis), inflammation of the muscle- or tendon insertions at adjacent bone (enthesitis), as well as raised red patches or various other expressions of psoriasis on the skin. Guselkumab (TREMFYA) is a fully human immunoglobulin G1 lambda (IgG1) monoclonal antibody (mAb) that binds to the p19 subunit of human interleukin (IL) 23 with high specificity and affinity, blocking IL-23 binding. Binding of guselkumab to the IL-23p19 subunit blocks the subsequent binding of extracellular IL-23 to the cell surface IL-23 receptor, inhibiting IL-23 specific intracellular signaling and subsequent activation and cytokine production. Participants with confirmed diagnosis of PsA who are starting guselkumab or any marketed interleukin-17 inhibitor (IL-17i) as a first, second, third, or fourth line of PsA biologic therapy per standard clinical practice will be enrolled in the main study. The aim of main study is to document the use of guselkumab and approved IL-17i therapies in routine clinical practice in patients with PsA who are starting guselkumab or an IL-17i as a first, second, third, or fourth line of biologic disease-modifying antirheumatic drugs (bDMARD) therapy. The overall duration of the main study, including recruitment and follow-up, is expected to be about 6 years. Participants who are starting guselkumab or an IL-17i treatment per routine clinical practice in the main study, and who meet the selection criteria for both the main study and substudy, will be consecutively offered entry into the substudy (a select number) at the time of enrollment into the main study. The substudy aims to collect additional data, continuously or with increased frequency, on the impact of guselkumab or IL-17i on patient mood, physical activity, sleep disturbance, disease symptoms, and health-related quality-of-life (HRQoL). Total duration of the substudy will be approximately 26-30 weeks consisting of a pre-treatment period of up to 14 days before the first dose of guselkumab or IL-17i in the main study and a 24-week (plus [+] up to 4 weeks follow-up) observation period.

ELIGIBILITY:
Inclusion Criteria:

Main study:

* Have a confirmed diagnosis of PsA as determined by a rheumatologist with reference to Classification criteria for Psoriatic Arthritis (CASPAR)
* Start guselkumab or any approved interleukin-17 inhibitor (IL-17i) as a first, second, third, or fourth line of biologic disease-modifying antirheumatic drugs (bDMARD) therapy for the indication of PsA as part of standard clinical practice (according to local label, local regulations, and/or reimbursement requirements) at the time of enrollment into the observational study or within a maximum of 2 months after the initial baseline visit or after repeated baseline data collection
* Sign a participation agreement/Informed consent form (ICF) allowing data collection and source data verification in accordance with local requirements
* Able to read, understand, and intend to comply with completion of all Electronic patient-reported outcome (ePRO) instruments
* The treatment decision must be taken by the participating rheumatologist prior to, and independently of the participant's inclusion into the study, following clinical practice in accordance with local and overarching guidelines and local regulations

Substudy:

* Must sign the substudy ICF allowing data collection in accordance with local requirements
* Is scheduled to receive guselkumab or IL-17i, per routine clinical practice, in the main study
* Currently using or is willing to use wearables and/or commercial applications to track their disease within the course of their normal daily activities

Exclusion Criteria:

Main study:

* Start guselkumab or an IL-17i therapy as fifth or further line of biologic treatment
* Have already taken a specific IL-17i or IL-23i treatment and are planning on re-taking that specific treatment again
* Unwilling or unable to participate in long-term data collection
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 30 days before the start of the study (that is, signing of informed consent)
* Currently enrolled in any interventional study or any Janssen-sponsored observational clinical study (contemporary participation into observational studies or registries not sponsored by Janssen is acceptable)

Substudy:

* Have an insufficient command of language to interact effectively with the smartphone application, in the opinion of the investigator at each site
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient (example, compromise the well-being) or that could prevent, limit, or confound assessment
* Unwilling or unable to comply with substudy assessments

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of participants initially treated for Psoriatic Arthritis (PsA) with guselkumab or interleukin-17 inhibitor (IL-17i) per routine clinical practice in accordance with clinical guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 1314 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
The Start and Stop Date of Guselkumab, as Applicable, For Each Participant | Up to 39 months
  The start and stop date, (first and last administration date, respectively) of guselkumab, as applicable, for each participant will be collected to document treatment persistence.
The Start and Stop Date of Interleukin-17 Inhibitor (IL-17i), as Applicable, For Each Participant | Up to 39 months
  The start and stop date (first and last administration date respectively) of IL-17i, as applicable, for each participant will be collected to document treatment persistence.

SECONDARY OUTCOMES:
Change from Baseline in 66 and 68 Joint Counts for Swelling and Tenderness, Respectively | Baseline up to 39 months
  Change from baseline in 66 and 68 joint counts for swelling and tenderness, respectively will be reported. Joints assessed include the distal interphalangeal, proximal interphalangeal, and metacarpophalangeal joints of the hands; the wrist, elbow, shoulder, acromioclavicular, sternoclavicular, temporomandibular, hip (excluded for swelling), knee, ankle, and midtarsal joints; and the metatarsophalangeal and proximal interphalangeal joints of the feet.
Change from Baseline in Rheumatologist's Global Assessment of Disease Activity-Psoriatic Arthritis (PGA-PsA) | Baseline up to 39 months
  The PGA-PsA will be documented using a Visual Analogue Scale (VAS) that ranges from "no PsA activity" (0 Millimeter [mm]) to "extremely active PsA" (100 mm).
Change from Baseline in Assessment of Dactylitis | Baseline up to 39 months
  The presence of and total number of digits of the hands and feet (that is, 0 to 20) with dactylitis will be documented.
Change from Baseline in Assessment of Enthesitis using Leeds Enthesitis Index (LEI) | Baseline up to 39 months
  The presence and a score of enthesitis will be documented using the LEI to evaluate the presence (score of 1) or absence (score of 0) of pain by applying local pressure to the following entheses: the lateral epicondyles (left and right), medial femoral condyles (left and right), and Achilles tendon insertions (left and right).
Change from Baseline in Nail Involvement | Baseline up to 39 months
  Nail involvement will be documented by recording the total number of nails of the hands and feet (that is, 0 to 20) with psoriatic nail changes.
Change from Baseline in Body Surface Area (BSA) Psoriasis (PSO) Skin Involvement | Baseline up to 39 months
  The BSA score indicates the surface area of the participant's body effected by psoriasis.
Change from Baseline in C-reactive Protein (CRP) | Baseline up to 39 months
  Change from baseline in CRP will be reported.
Change from Baseline in Minimal Disease Activity (MDA)/ Very Low Disease Activity (VLDA) | Baseline up to 39 months
  Change from Baseline in MDA/VLDA will be reported.
Change from Baseline in Clinical Disease Activity Index for Psoriatic Arthritis (cDAPSA/DAPSA) | Baseline up to 39 months
  DAPSA assesses the joint domain of PsA and is derived from the sum of the following components: Participant's assessment of pain on VAS (in centimeters), Participant's Global Assessment of Disease Activity on VAS (in centimeters), 66 and 68 joint counts for swelling and tenderness, respectively.
Response as a Measure of Clinical Improvement in cDAPSA/DAPSA | Up to 39 months
  Response is defined as a clinical improvement in cDAPSA/DAPSA. DAPSA assesses the joint domain of PsA and is derived from the sum of the following components: Participant's assessment of pain on VAS (in centimeters), Participant's Global Assessment of Disease Activity on VAS (in centimeters), 66 and 68 joint counts for swelling and tenderness, respectively.
Start and Stop Dates of All Treatments and the Sequence of Treatment Lines | Up to 39 months
  Start and stop dates of all treatments and the sequence of treatment lines will be reported.
Percentage of Participants with Adverse Events (AEs) | Up to 39 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
BSA PSO Skin Involvement | Up to 39 months
  The BSA score indicates the surface area of the participant's body affected by psoriasis.
Rheumatic Disease Comorbidity Index | Up to 39 months
  Number of comorbid medical conditions of the study participants for the Rheumatic Disease Comorbidity Index will be reported.
Change from Baseline in Fibromyalgia Rapid Screening Tool (FiRST) | Baseline up to 6 months
  FiRST will be used to help determine whether participants have chronic widespread pain or fibromyalgia syndrome at entry into the study. The FiRST is a validated questionnaire consisting of a combination of 6 items that can detect chronic widespread pain.
Change from Baseline in European Quality of Life (EuroQoL) 5-Dimensions 5-Levels Questionnaire (EQ-5D-5L) | Baseline up to 39 months
  The EQ-5D-5L is a standardized instrument for use as a measure of health outcome, primarily designed for self-completion by respondents. The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of the 5 dimensions is divided into 5 levels of perceived problems, where Level 1: no problem, Level 2: slight problems, Level 3: moderate problems, Level 4: severe problems and Level 5: extreme problems.
Change from Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) | Baseline up to 39 months
  The functional status of the participants will be assessed by the HAQ-DI. This 20-question self-administered instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area.
Change from Baseline in Psoriatic Arthritis Impact of Disease-12 (PsAID-12) | Baseline up to 39 months
  PsAID-12 is a validated, self-administered questionnaire that assesses the impact of PsA on participants' lives. It consists of 12 questions, each answered using a numerical rating scale. Questions related to pain, skin problems, work and/or leisure activities, discomfort, embarrassment and/or shame, social participation, and anger, fear, and uncertainty, and depression are scored from 0 (none) to 10 (extreme), functional capacity and sleep disturbance are scored from 0 (no difficulty) to 10 (extreme difficulty) and coping is scored from 0 (very well) to 10 (very poorly).
Change from Baseline in Patient Global Disease Activity Visual Analog Scale (VAS) Scores | Baseline up to 39 months
  The Patient Global Disease Activity VAS is a self-administered assessment with scores ranging from "very well" (0 mm) to "very poor" (100 mm) that assesses disease activity over the past week.
Change from Baseline in Pain VAS Score | Baseline up to 39 months
  The pain VAS is a self-administered assessment of average pain during the past week. The scale ranges from "no pain" (0 mm) to "the worst possible pain" (100 mm).
Change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline up to 39 months
  BASDAI consists of a 1 through 10 scale (1 being no problem and 10 being the worst problem) which is used to answer 6 questions pertaining to the 5 major symptoms of ankylosing spondylitis: fatigue, spinal pain, joint pain/swelling, areas of localized tenderness (also called enthesitis, or inflammation of tendons and ligaments), morning stiffness duration, morning stiffness severity.
Change from Baseline in Ankylosing Spondylitis Disease Activity Score - C-reactive protein (ASDAS-CRP) | Baseline up to 39 months
  The ASDAS-CRP is a composite of 5 disease activity variables with only partial overlap. The 4 self-reported items included in this index are back pain (VAS), duration of morning stiffness, peripheral pain/swelling, and participant global assessment of disease activity; these are combined with the CRP value.
Change from Baseline in Dermatology Life Quality Index (DLQI) | Baseline up to 39 months
  The DLQI is a dermatology-specific, validated, 10-question quality of life instrument used to measure the impact of skin disease on the quality of life of an affected person. Each question will address how much the participant's skin problem has affected their life and is scored as: 3 = very much, 2 = a lot, 1 = a little, 0 = not at all, or not relevant.
Change from Baseline in Patient Acceptable Symptom State (PASS) | Baseline up to 39 months
  The PASS measures the level of symptoms beyond which participants consider themselves well. The PASS addresses the concepts of low disease activity, partial remission in symptoms, and well-being.
Change from Baseline in Work Productivity and Activity Impairment Questionnaire: Psoriatic Arthritis (WPAI: PsA) | Baseline up to 39 months
  The WPAI: PsA is a validated, self-administered questionnaire that assesses work and activity impairment during the past 7 days. The WPAI: PsA produces 4 types of scores: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment. The WPAI: PsA outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, that is, worse outcomes.
Change from Baseline in Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9) | Baseline up to 39 months
  TSQM-9 is a 9-item, validated, self-administered instrument used to assess participant's satisfaction with medication. The three domains assessed are effectiveness, convenience, and side effects of the medication.
Number of Participants Switching or Stopping Treatment | Up to 39 months
  Number of Participants switching or stopping treatment (including reasons for discontinuation) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (154):
- Argentina (5):
  - OMI, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital J. M. Ramos Mejía, Buenos Aires
  - Hospital Cordoba, Córdoba
  - MR Medicina Reumatologica, San Fernando
- Australia (3):
  - The Queen Elizabeth Hospital, Adelaide
  - Footscray Hospital, Western Health, Footscray
  - Royal North Shore Hospital, St Leonards
- Austria (4):
  - LKH-Univ. Klinikum Graz, Graz
  - Kepler Universitatsklinikum GmbH, Linz
  - Medizinische Universitaet Wien, Vienna
  - Evang. Krankenhaus Gemein. Betriebgesm. Mbh, Vienna
- Belgium (5):
  - AZ Sint-Jan, Bruges
  - Hopital Erasme, Brussels
  - Reumaclinic Genk-Hasselt, Genk
  - UZ Leuven, Leuven
  - CHU de Liège - Domaine Universitaire du Sart Tilman, Liège
- Canada (16):
  - Artus Health Centre, Vancouver, British Columbia
  - Manitoba Clinic, Winnipeg, Manitoba
  - Dr. Juris Lazovskis Incorporated, Coxheath, Nova Scotia
  - Private Practice - Dr. Pauline Boulos, Dundas, Ontario
  - Markham Rheumatology Hub, Markham, Ontario
  - Brandusa Florica Medicine Professional Corporation, Mississauga, Ontario
  - The Waterside Clinic, Orillia, Ontario
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Dr Sabeen Anwar Medicine Professional Corporation, Windsor, Ontario
  - CIUSSS de l Est de l Ile de Montreal Installation Hopital Maisonneuve Rosemont, Montreal, Quebec
  - G R M O Groupe de recherche en maladies osseuses Inc, Québec, Quebec
  - Centre de sante et services sociaux (CSSS) de Rimouski-Neigette - Hopital regional - Rimouski, Rimouski, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Centre de Recherche Musculo Squelettique, Trois-Rivières, Quebec
  - Community Rheumatology Care, Saskatoon, Saskatchewan
  - Rheumatology Associates of Saskatoon, Saskatoon, Saskatchewan
- Colombia (5):
  - BIOMAB, Bogotá
  - Servimed S A S, Bucaramanga
  - Clinisalud del Sur, Medellín
  - Clinica Vascular las Americas, Medellín
  - Funcentra, Montería
- France (16):
  - Hôpital Avicenne, Bobigny
  - Centre Hospitalier de Cholet, Cholet
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier Universitaire(CHU) - Hopital Henri Mondor, Créteil
  - CHU Grenoble, Échirolles
  - CHRU HOPITAL ROGER SALENGRO Consultation Appareil locomoteur, Lille
  - Centre Orthopedique Santy, Lyon
  - Clinique de l'Infirmerie Protestante de Lyon, Lyon
  - Hôpital Saint Roch, Nice
  - CHR Orléans - Nouvel Hôpital Orléans La Source, Orléans
  - Hôpital Lariboisière - Centre Viggo Petersen, Paris
  - Hopital Saint-Antoine, Paris
  - Hôpital Bichat, Paris
  - Hôpital Pitié-Salpétrière, Paris
  - CHRU Hôpital de Hautepierre, Strasbourg
  - Hopital Purpan, Toulouse
- Germany (19):
  - Praxis für Rheumatologie, Amberg
  - Rheuma-Praxis Bayreuth, Bayreuth
  - Rheumatologische Schwerpunktpraxis, Berlin
  - Krankenhaus Porz am Rhein, Cologne
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Service Rheuma Erfurt, Erfurt
  - Universitatsklinikum Frankfurt, Frankfurt
  - Rheumapraxis Dr. Liebhaber, Halle
  - Praxis fur Klinische Studien und Praxis fur Orthopadie, Hamburg
  - Rheumatologie im Struenseehaus, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - Rheumatologische Praxis, Leipzig
  - Rheumatologische Praxis, Magdeburg
  - Praxiszentrum St. Bonifatius, München
  - Praxis Thilo Klopsch, Neubrandenburg
  - Knappschaftsklinikum Saar GmbH Klinik für Rheumatologie, Püttlingen
  - Rheumazentrum Ratingen, Ratingen
  - Rheumatologisch-immunologische Arztpraxis, Templin
  - Immunologisches Zentrum Vogelsang-Gommern GmbH, Vogelsang-Gommern
- Greece (9):
  - Evangelismos General Hospital of Athens, Athens
  - Athens Navy Hospital, Athens
  - General Hospital 'Gennimatas', Athens
  - Hippokration General Hospital of Athens, B' Internal Medicine Clinic,, Athens
  - Laiko General Hospital of Athens, Athens
  - University Hospital of Ioannina, Ioannina
  - 'Agios Andreas' General Hospital of Patras, Pátrai
  - University General Hospital of Rio Patras, Pátrai
  - Ippokrateio Hospital, Thessaloniki
- Italy (14):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Ospedale Regionale Cardarelli-Università degli Studi del Mol, Campobasso
  - Universita della Magna grecia, Catanzaro
  - AOU Careggi, Florence
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Seconda Univesità degli Studi di Napoli, AOU, Napoli
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale San Carlo Di Potenza - Azienda Ospedaliera Regionale, Potenza
  - Universita Cattolica del Sacro Cuore, Rome
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliero Universitaria S.Maria Della Misericordia, Udine
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (6):
  - Kita-harima Medical Center, Hyōgo
  - Toho University Medical Center, Ohashi Hospital, Meguro-ku
  - Osaka Metropolitan University Hospital, Osaka
  - Public Interest Incorporated Foundation Nipoon Life Saiseikai Nippon Life Hospital, Osaka
  - Hokkaido University Hospital, Sapporo
  - Kyorin University Hospital, Tokyo
- Mexico (3):
  - Medical Care & Research SA de CV, Mérida
  - Consultorio de Reumatologia, México
  - Hospital Puerta de Hierro, Zapopan
- Netherlands (4):
  - Academisch Medisch Centrum Universiteit van Amsterdam, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Universitair Medisch Centrum Groningen, Groningen
  - Elkerliek Ziekenhuis, Helmond
- Russia (4):
  - SBEU HPE Kemerovo State Medical Academy, Kemerovo
  - Bakoulev Scientific Center For Cardiovascular Surgery Rams, Moscow
  - FGBU Research Institute of Rheumatology named V.A.Nasonova, Moscow
  - City Hospital #3, Tomsk
- South Korea (4):
  - Soonchunhyang University Cheonan Hospital, Cheonan-si
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
- Spain (12):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Punta de Europa, Algeciras / Cadiz
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. de Basurto, Bilbao
  - Hosp Reina Sofia, Córdoba
  - Complejo hospitalario de Granada, Granada
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. de Getafe, Madrid
  - Hosp. Univ. Central de Asturias, Oviedo
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Virgen Del Rocio, Seville
- Sweden (5):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Universitetssjukhuset i Lund, Lund
  - Universitetssjukhuset Orebro, Örebro
  - Akademiskt Specialistcentrum centrum för reumatologi, Stockholm
  - Akademiska Sjukhuset, Uppsala
- HFR Fribourg - Hôpital Cantonal, Fribourg, Switzerland
- Taiwan (3):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
- United Kingdom (16):
  - NHS Grampian - Aberdeen Royal Infirmary (ARI), Aberdeen
  - Nevill Hall Hospital, Abergavenny
  - University Hospital Monklands, Airdrie
  - Royal Free London NHS Foundation Trust Barnet Hospital, Barnet
  - Wolfson Centre Royal United Hospitals, Bath
  - Glasgow Royal Infirmary, Glasgow
  - Hull Royal Infirmary, Hull
  - Leeds Teaching Hospitals NHS Trust Chapel Allerton Hospital, Leeds
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - The Newcastle upon Tyne Hospitals NHS Trust - Freeman Hospit, Newcastle upon Tyne
  - Queen Alexandra Hospital, Portsmouth
  - Shirley Caldwell, Salford
  - Southampton General Hospital, Southampton
  - Haywood Hospital, Staffordshire
  - Stamford and Rutland hospital, Stamford
  - Wishaw General, Wishaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siebert S, Behrens F, Lubrano E, Martin N, Sharaf M, Contre C, Theander E, Queiro R, Zimmermann M, Gossec L. PsABIOnd Study and eDaily Substudy Design: Long-Term Effectiveness and Safety of Guselkumab and IL-17 Inhibitors in Routine Clinical Practice in Patients with Psoriatic Arthritis. Rheumatol Ther. 2023 Apr;10(2):489-505. doi: 10.1007/s40744-022-00518-w. Epub 2022 Dec 30. PMID 36585602